CLINICAL TRIAL: NCT04309253
Title: The Influence of Vascular Burden, Amyloid Plaque and Tau Protein in Patients With Vascular Cognitive Impairment and Dementia With Tauopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201800984A0
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Vascular Cognitive Impairment, Alzheimer's Disease, Fronto-temporal Dementia
Keywords: Vascular cognitive impairment, Alzheimer's disease, fronto-temporal dementia, amyloid plaque, tau protein
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: A. Group A: Patients with vascular cognitive impairment (VCI), n=80. B. Group B: Alzheimer's disease/mild cognitive impairment (MCI), n=80. C. Group C: Fronto-temporal dementia (FTD), n=30. D. Group D: Normal control, n=30. E. Group E: progressive supranuclear palsy(PSP), n=80.
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMPBB3 (Other): 1. Primary endpoint(s):
     A. To determine the distribution patterns of cerebral amyloid plaques and Tau protein among AD/MCI, VCI and FTP patients as well as normal controls.
  2. Secondary endpoints:
  A. To correlate vascular burden, [18F]AV45 and [18F]MNI-958(PMPBB3) retention with clinical presentation and cognitive performance among different groups of subjects B. To determine the impacts of vascular burden, [18F]AV45 and [18F]MNI-958(PMPBB3) retention changes on cognitive trajectory over the 18-month follow-up period.
  Interventions: Drug: PMPBB3; Drug: AV45
- AV45 (Other): 1. Primary endpoint(s):
     A. To determine the distribution patterns of cerebral amyloid plaques and Tau protein among AD/MCI, VCI and FTP patients as well as normal controls.
  2. Secondary endpoints:
  A. To correlate vascular burden, [18F]AV45 and [18F]MNI-958(PMPBB3) retention with clinical presentation and cognitive performance among different groups of subjects B. To determine the impacts of vascular burden, [18F]AV45 and [18F]MNI-958(PMPBB3) retention changes on cognitive trajectory over the 18-month follow-up period.
  Interventions: Drug: PMPBB3; Drug: AV45

INTERVENTIONS:
Drug: PMPBB3 — F-18 PMPBB3 PET Imaging
Drug: AV45 — F-18 AV45 PET Imaging

SUMMARY:
Background and objects Amyloid plaques and tau protein are the landmarks of neurodegeneration in Alzheimer's disease (AD). On the other hand, it is reported that cerebral ischemia may induce amyloid plaques and tau protein accumulation. However, it was difficult to in vivo disentangle the complex and dynamic interactions between AD pathophysiology and cerebral vascular injury during the post-stroke cognitive impairment development in the past. With the advent of novel radiotracers specific to cerebral amyloid plaques and tau protein, we aim to conduct a prospective multimodal neuroimaging cohort study to investigate the contribution of vascular injury, amyloid plaque and tau protein to cognitive impairment.

Subjects and methods The prospective project plans to recruit patients with vascular cognitive impairment (VCI) (Group A, n=80), Alzheimer's disease/mild cognitive impairment (MCI) (Group B, n = 120), fronto-temporal dementia (FTD) (Group C, n =30), and progressive supranuclear palsy (PSP) (Group E, n = 80). In addition, another 30 healthy people will be recruited as the control group (Group D, n=30). [18F]AV45 and [18F]MNI-958(PMPBB3) PET will be done for imaging cerebral amyloid plaque and tau protein distribution, brain MRI for obtaining structural and functional information, and neuropsychological tests for cognitive performance. Cognitive evaluation will be repeated 18 months after recruitment. In addition, APOE genotyping will be performed as well.

By obtaining the neuroimaging information, such as severity of white matter change and infarction, cortical and hippocampal atrophy, and SUVRs of [18F]AV-45 and [18F]MNI-958(PMPBB3) PET, the study will be able to investigate the composite influence of cerebrovascular disease and neurodegenerative pathology on the trajectory of cognitive impairment. Group comparisons will be performed using the Chi-square test, independent t test, Mann-Whitney U test, ANOVA test, and multiple linear regression, where appropriate.

Anticipation In this project, we will be able to explore the distribution patterns of amyloid plaque and tau protein among dementia patients with different etiologies, and also evaluate their influence on cognition

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for VCI (Group A, n=80)

   * Males or females with age >= 20 years old.
   * Patients fulfill the AHA/ASA criteria for vascular cognitive impairment.
   * Provision of signed informed consent from the subject and the subject's legally authorized representative or caregiver (if applicable).
   * The subject has an appropriate caregiver capable of accompanying the subject, if necessary.
2. Inclusion criteria for AD / MCI (Group B, n=120)

   * Males or females with age >= 20 years old.
   * Patients fulfill the National Institute on Aging (NIA) - Alzheimer's Association Diagnostic Guidelines.
   * Provision of signed informed consent from the subject and the subject's legally authorized representative or caregiver (if applicable).
   * The subject has an appropriate caregiver capable of accompanying the subject, if necessary.
3. Inclusion criteria for FTD (Group C, n=30)

   * Males or females with age >= 20 years old.
   * Patients fulfill the criteria of probable FTD.
   * Provision of signed informed consent from the subject and the subject's legally authorized representative or caregiver (if applicable).
   * The subject has an appropriate caregiver capable of accompanying the subject, if necessary.
4. Inclusion criteria for normal control (Group D, n=30)

   * Males or females with age >= 20 years old.
   * Provision of signed informed consent.
5. Inclusion criteria for PSP (Group E, n=80)

   * Males or females with age >= 20 years old
   * Patients fulfill the 2017 Movement Disorder Society criteria of PSP.
   * Provision of signed informed consent from the subject and the subject's legally authorized representative or caregiver (if applicable)
   * The subject has an appropriate caregiver capable of accompanying the subject, if necessary.

Exclusion Criteria:

* Life expectancy less than 1 year.
* Clinically significant abnormal laboratory values (such as AST/ALT >= 3X of upper normal limits).
* Clinically significant or unstable medical or psychiatric illness.
* Epilepsy history.
* Cognitive impairment resulting from trauma or brain damage.
* Substance abuse or alcoholism in the past 3 months.
* Stroke history within the recent 3 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-09-21 (Actual); Primary Completion 2024-05-18 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
The Clinical Dementia Rating-Sum of Boxes (CDR-SB) change score | through study completion, an average of 1.5 year
  The Clinical Dementia Rating-Sum of Boxes (CDR-SB) change score between baseline and 18-month follow-up will be calculated for primary endpoint determination. Two-sample independent t-test will be performed to compare the CDR-SB change score between patients positive and negative for tau protein accumulation. Patients will be stratified into tau-positive and tau-negative groups, and the presentations of their cognitive state will be recorded at the 18-month follow-up visit.
Chi-square test will be performed to analyze dementia conversion rate. | through study completion, an average of 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Huang Kuo-Lun, M.D., Study Chair — Stroke Section, Department of Neurology, Chang-Gung memorial Hospital
Locations (1):
- Department of Neurology, Chang-Gung memorial Hospital, Taoyuan District, Guishan, Taiwan